CLINICAL TRIAL: NCT03228602
Title: Gustatory Evoked Potentials and Cerebral Control of Food Intake in Obese Subjects
Brief Title: Impaired Gustatory Sensory Perception in Obese and Obese Diabetic Persons
Acronym: PEGASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JACQUIN PEGASE 2016
Record Dates: First submitted 2017-06-26; First posted 2017-07-25 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- healthy subjects (Active Comparator)
  Interventions: Other: Recording of GEP (Gustatory Evoked Potentials)
- obese (Experimental)
  Interventions: Other: Recording of GEP (Gustatory Evoked Potentials)
- obese diabetic (Experimental)
  Interventions: Other: Recording of GEP (Gustatory Evoked Potentials)
- obese diabetic who are going to be operated on (Experimental): 25 of a sleeve gastrectomy and 25 of a Y gastric bypass
  Interventions: Other: Recording of GEP (Gustatory Evoked Potentials)

INTERVENTIONS:
Other: Recording of GEP (Gustatory Evoked Potentials) — record cerebral activity thanks to electrodes placed on the head and fixed with a painless, harmless adhesive paste and linked to a computer equipped with specific software to interpret the signals obtained. The collection of data for the electric signal takes 20 minutes.

SUMMARY:
The aim of the study is to compare several parameters in three distinct groups of subjects: persons with obesity, persons with obesity and diabetes and persons with neither obesity nor diabetes:

* the electrical activity in response to a sweet solution, measured before and after a standard meal, using gustatory evoked potentials (recording explained below)
* blood hormone levels related to weight gain (insulin, dopamine, ghrelin, leptin: measured in blood samples)
* levels of activity and quantity of an enzyme present in the saliva, amylase, which is able to break down ingested starch into several molecules of glucose.

All of these parameters will be correlated to determine whether the results are different in the 3 groups of subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written consent
* Patients over 18 years old
* Body Mass Index (BMI) <25 kg/m² for healthy volunteers and BMI≥30 kg/m² for obese subjects
* Patients with type 2 diabetes for the group "obese diabetic subjects"

Exclusion Criteria:

* Patients under guardianship
* Patients without health insurance cover
* Pregnant or breast-feeding women
* Active smokers
* Subjects with type 2 diabetes for the " healthy subjects " and " obese subjects ", subjects with type 1 diabetes for all groups
* Subjects who do not speak French
* Treatment that interferes with taste or acts on the central nervous system
* Anti-diabetic treatment with GLP-1 analogues (Glucagon-like peptide 1) or SGLT2 (sodium-glucose cotransporter type 2)
* Known hypersensitivity to the foods proposed in the study, or the paste used to fix the electrodes, or to paraffin wax or to the products tested (sucrose, glucose or starch for the gustatory evoked potentials and triangular tests)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Amplitude of the gustatory evoked potential | Up to 10 days
Latency of the gustatory evoked potential | Up to 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France